CLINICAL TRIAL: NCT03161795
Title: Addressing the Risks of Long-Term Opioid Therapy in Chronic Noncancer Pain: A National, Multicenter, and Observational Cross-sectional Study in South Korea
Brief Title: Addressing the Risks of Long-Term Opioid Therapy in Chronic Noncancer Pain
Status: Completed | Type: Observational
Sponsor: Seoul National University (Other)
Collaborators: Seoul National University Bundang Hospital (Other); Korea University Guro Hospital (Other); Ewha Womans University (Other); Ajou University School of Medicine (Other); Konkuk University Hospital (Other); Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other); Seoul St. Mary's Hospital (Other)
Responsible Party: Principal Investigator, Jeeyoun Moon, Clinical Associate Professor, Seoul National University
Other Study IDs: 1702-020-829
Record Dates: First submitted 2017-05-16; First posted 2017-05-22 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Chronic Noncancer Pain; Opioid-Related Disorders
Keywords: Chemical coping; Long-term opioid therapy; Risk factors; Predictive tools; Frequency
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
PURPOSE: Assess the risks of long-term opioid therapy, especially opioid use disorders such as opioid-related chemical coping in chronic noncancer pain patients.

Pain, particularly chronic pain, is a major threat to the quality of life worldwide and will become more so as the average age increases. Currently, over 30% of the world's population is known to have chronic pain. Among a plethora of treatment options, opioid agonists is one of treatment options for moderate to severe chronic pain. Although its consumption has increased during the last two decades,3 it remains below the requirements in most regions, including the Asian countries. In South Korea (S. Korea), opioid consumption for medical purposes in 2015 was still below average, ranked 43rd globally and 30th among 35 Organisation for Economic Co-operation and Development (OECD) countries (55 mg/capita in S. Korea vs. 258 mg/capita in an average of OECD countries). Conversely, in countries with high opioid consumption such as the United States of America (US), drug overdose deaths (the majority involving an opioid) have nearly quadrupled since 1999.

The up to date literature on opioid use disorder (OUD) is characterized by great variability of definitions, measurements, demographics, and opioid use duration. Moreover, an overwhelming majority of the studies took place in the US, the country with the highest opioid consumption and a current opioid crisis. Additionally, stringent restrictions and regulations to prevent OUD may result in inadequate pain control and insufficient opioid therapy, especially in countries with relatively low-moderate opioid consumption rates. Therefore, in compliance with growth in medical opioid use and the lack of studies in countries with low-moderate opioid consumption, it is necessary to determine the occurrence of OUD in chronic noncancer pain (CNCP) patients receiving long-term opioid therapy (LtOT).

In this study, we will perform a national, multicenter, observational cross-sectional study to address the current status of opioid treatment for CNCP in S. Korea, a country with moderate opioid consumption. The ultimate aims of this study are to estimate the frequency of OUD such as OrCC, to evaluate the functional and psychiatric characteristics of patients, and to determine the risk factors associated with OUD in CNCP patients receiving LtOT.

DETAILED DESCRIPTION:
Chronic pain is a devastating disease often treated inadequately. More than 30 percent of the world population suffers from chronic pain. Among a plethora of treatment options, opioid agonists is one of treatment options for moderate to severe chronic pain. Although its consumption has increased during the last two decades, it remains below the requirements in most regions, including the Asian countries. In South Korea (S. Korea), opioid consumption for medical purposes in 2015 was still below average, ranked 43rd globally and 30th among 35 Organisation for Economic Co-operation and Development (OECD) countries (55 mg/capita in S. Korea vs. 258 mg/capita in an average of OECD countries). However, it is remarkable that the opioid consumption in S. Korea has increased 5-6 times since 2005 (10 mg/capita), ranking 3rd among Asian countries, preceded only by Vietnam (62 mg/capita) and Malaysia (60 mg/capita).

One of the reluctant factors to prescribe opioids is induced reward responses, resulting in opioid use disorders (OUD). Particularly, in chronic noncancer pain (CNCP), concerns regarding drug dependence in the long-term opioid therapy (LtOT) remain its use controversial. The spectrum of OUD in CNCP patients is wide and varies from misuse without a compliant intake to addiction with a severe aberrant consumption. Between the extremes, opioid-related chemical coping (OrCC) may lie in a middle ground group, characterized by an inappropriate use of opioids to cope with emotional distress. Although, OrCC is a terminology first used in cancer patients, a recent study found a high correlation between the reports of aberrant medication-taking behavior by experienced providers and chemical coping by CNCP patients.

OrCC should be distinguished from psychologic addiction, a neurobiological disease that corresponds with the most severe substance-use disorder referring to neuroplasticity and a substantial loss of self-control. All addicts are eventually chemical copers, but not all chemical copers are addicts. A better understanding of this intermediate status may be crucial to prompt to identify the risk of severe OUD and re-direct their management to avoid unnecessary opioid toxicity and achieve adequate pain control. However, studies to measure OrCC are scarce and the evidence of OUD in CNCP in countries with relatively low opioid consumption is practically unavailable.

The up to date literature on OUD is characterized by great variability of definitions, measurements, demographics, and opioid use duration. Moreover, an overwhelming majority of the studies took place in the United Stated of America (US), the country with the highest opioid consumption and a current opioid crisis. Despite their over-consumption, however, studies in those countries showed that CNCP is still undertreated and even suggested that OUD might not be related to the prescription to pain patients. From a different angle, stringent restrictions and regulations to prevent OUD may result in inadequate pain control and insufficient opioid therapy, especially in countries with relatively low- moderate opioid consumption rates. Therefore, to strike a balance when treating pain with opioids, it is indispensable to determine the characteristics of OUD in CNCP patients with LtOT in countries with low-moderate opioid consumption. Moreover, in S. Korea there are not available statistics regarding the OUD occurrence in CNCP patients and national guidelines on LtOT in CNCP have not been developed.

In this study, we will perform a national, multicenter, observational cross-sectional study to address the current status of opioid treatment and OUD for CNCP in S. Korea, a country with moderate opioid consumption since 2010. The availability of up-to-date data on OUD is necessary for the development of national guidelines to prevent severe harms of opioids, enhance patients and physicians' satisfaction, potentiate opioid's benefits, and guaranty adequate pain control in the CNCP population. The ultimate aims of this study are to estimate the frequency of OUD (such as OrCC), to evaluate the patient's functional and psychiatric characteristics, and to determine the risk factors associated with OUD in CNCP patients receiving LtOT. The results of this study will help to seize the occurrence of OUD in countries with low-moderate opioid consumption thus it will approach the real risk effect of LtOT in CNCP.

ELIGIBILITY:
Inclusion criteria were as follows: 1) patients at age equal or greater than 18 years; 2) patients with a diagnosis of chronic pain defined by the American Chronic Pain Association (ACPA) as an ongoing or recurrent pain, lasting beyond the usual course of acute illness or injury or more than 3 months, and which adversely affected the individuals' well-being; 3) patients with CNCP with opioid medication for treatment and/or control of chronic pain; 4) patients who were receiving long-term opioid therapy defined as the use of opioids on most days for a period of time greater than 3 months; and 5) patients who complete the screening tools and questionnaires evaluated in the study.

Exclusion criteria were as follows: 1) patients with diagnosis and/or ongoing cancer treatment or palliative or receiving end-of-life care; 2) patients younger than 18 years of age; 3) patients without current opioid therapy for the treatment and/or control of chronic pain; 4) patients with chronic pain that received opioid therapy intermittently or for less than 3 months; 5) serious systemic diseases (Myasthenia Gravis, decreased lung function, severe liver problems, severe renal impairment, shock, hypo- or hyperpotassemia) or psychiatric disorders (schizophrenia and acute anxiety) that compromise the patients safety or the completion of the survey; or 6) patients with intellectual impairment to answer the tools and questionnaires evaluated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study was open-labeled, national, multicenter, observational, cohort study conducted at 8 Tertiary hospitals located in South Korea. The study population were patients with chronic noncancer pain receiving long-term opioid therapy and attending the outpatient pain clinic of any of the participant hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 258 (Actual)
Dates: Start 2017-04-25 (Actual); Primary Completion 2018-01-19 (Actual); Study Completion 2018-03-12 (Actual)

PRIMARY OUTCOMES:
Frequency of opioid-related chemical coping | The assessment took place during a routine outpatient clinic 1 day visit. The presence of chemical coping was evaluated by pain specialist through the questionnaire immediately after the routine visit of each patient.
  Prevalence of chemical coping with opioids in the study population by the pain specialists participating in the study through a questionnaire that contained the per-protocol definition of chemical coping and seven different aberrant behaviors related to chemical coping proposed by a panel of experts. One or more affirmative answers were considered as "positive"

SECONDARY OUTCOMES:
Sociodemographic characteristics of chronic noncancer pain patients using long-term opioid therapy | The data was collected from the start of the study up to 3 months after finishing recruitment. The NRS was assessed in each patient during the routine visit with a pain specialist.
  Patients' demographic data (sex, age, ethnicity, body mass index, marital status, education, and employment status), pain characteristics [duration, intensity using an 11-pointed numerical rating pain scale (NRS) score ranged from 0 (no pain) to 10 (pain as bad as you can imagine), etiology, location, and type of pain such as nociceptive, neuropathic, functional pain syndrome (fibromyalgia, temporomandibular disorder, etc.), and mixed, co-morbid psychiatric disease, substance abuse history, secondary morbid gain, ongoing litigation, history of taken prescription drugs with alcohol, and suicidal ideation] were collected.
Characteristic of opioid's use in chronic noncancer pain in South Korea | The data was collected from the start of the study up to 3 months after finishing recruitment.
  Opioid information including duration of administration, opioid types (long-acting vs. short-acting), route of administration (oral, transdermal, mucosal, or intravenous), Morphine Equivalent Daily Dosage (MEDD, mg/day), the initial prescriber, number of visits per year to an opioid prescriber, and history of Emergency room (ER) visits seeking for opioids, as well as concomitant use of benzodiazepines and other medication such as antidepressants, anticonvulsants, and/or topical agents were obtained.
Risk factors associated to long-term opioid therapy and opioid-related chemical coping | The patients answered to the questionnaires and tools before a routine 1 day visit. Each patient finished the evaluation on the same day of the visit. The record of answers will take place from the start to the finish of recruitment.
  The assessment was conducted through a survey in the outpatient setting of each pain clinic. The survey contained a number of questionnaires including 1) the Cut, Annoyed, Guilty, Eye-opener - Adapted to Include Drugs (CAGE-AID); 2) the Brief Pain Inventory-Short Form (BPI-SF); 3) Pain Catastrophizing Scale; 4) Hospital Anxiety and Depression Scale (HADS); 5) Insomnia Severity Index (ISI); 6) Korean Instrumental Activities of Daily Living Scale (K-IADL); 7) Korean-Connor-Davidson Resilience Scale (K-CD-RISC); and 8) Patient Global Impression of Change Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Jee Y Moon, MD, PhD, Study Director — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Relieving Pain in America: A Blueprint for Transforming Prevention, Care, Education, and Research. Mil Med. 2016 May;181(5):397-9. doi: 10.7205/MILMED-D-16-00012. No abstract available. PMID 27136641
- [Background] Kaplan JA, Richards-Waugh LL, Bailey KM, Kraner JC. Epidemic: fatal pharmaceutical abuse in West Virginia 1991-2008. W V Med J. 2010;106(4 Spec No):88-90. No abstract available. PMID 21932761
- [Background] Krnic D, Anic-Matic A, Dosenovic S, Draganic P, Zezelic S, Puljak L. National consumption of opioid and nonopioid analgesics in Croatia: 2007-2013. Ther Clin Risk Manag. 2015 Aug 28;11:1305-14. doi: 10.2147/TCRM.S86226. eCollection 2015. PMID 26357478
- [Background] Seya MJ, Gelders SF, Achara OU, Milani B, Scholten WK. A first comparison between the consumption of and the need for opioid analgesics at country, regional, and global levels. J Pain Palliat Care Pharmacother. 2011;25(1):6-18. doi: 10.3109/15360288.2010.536307. PMID 21426212
- [Background] Duthey B, Scholten W. Adequacy of opioid analgesic consumption at country, global, and regional levels in 2010, its relationship with development level, and changes compared with 2006. J Pain Symptom Manage. 2014 Feb;47(2):283-97. doi: 10.1016/j.jpainsymman.2013.03.015. Epub 2013 Jul 17. PMID 23870413
- [Background] Chung SS, Park CK, Cho KJ, Choi KH, Kim JH, Kim SB, Kuh SU, Lee JC, Lee JH, Lee KY, Lee SH, Moon SH, Park SY, Shim JH, Son BC, Yoon MH, Park HJ. A Nationwide Retrospective Study of Opioid Management Patterns in 2,468 Patients with Spinal Pain in Korea. Asian Spine J. 2016 Dec;10(6):1122-1131. doi: 10.4184/asj.2016.10.6.1122. Epub 2016 Dec 8. PMID 27994790
- [Background] Centers For Disease Control And Prevention Public Health Service U S Department Of Health And Human Services. Guideline for Prescribing Opioids for Chronic Pain. J Pain Palliat Care Pharmacother. 2016 Jun;30(2):138-40. doi: 10.3109/15360288.2016.1173761. PMID 27301691
- [Background] Breivik H, Cherny N, Collett B, de Conno F, Filbet M, Foubert AJ, Cohen R, Dow L. Cancer-related pain: a pan-European survey of prevalence, treatment, and patient attitudes. Ann Oncol. 2009 Aug;20(8):1420-33. doi: 10.1093/annonc/mdp001. Epub 2009 Feb 24. PMID 19244085
- [Background] O'Brien T, Christrup LL, Drewes AM, Fallon MT, Kress HG, McQuay HJ, Mikus G, Morlion BJ, Perez-Cajaraville J, Pogatzki-Zahn E, Varrassi G, Wells JC. European Pain Federation position paper on appropriate opioid use in chronic pain management. Eur J Pain. 2017 Jan;21(1):3-19. doi: 10.1002/ejp.970. PMID 27991730
- [Background] Kwon JH, Hui D, Bruera E. A Pilot Study To Define Chemical Coping in Cancer Patients Using the Delphi Method. J Palliat Med. 2015 Aug;18(8):703-6. doi: 10.1089/jpm.2014.0446. Epub 2015 Apr 29. PMID 25922879
- [Background] Del Fabbro E. Assessment and management of chemical coping in patients with cancer. J Clin Oncol. 2014 Jun 1;32(16):1734-8. doi: 10.1200/JCO.2013.52.5170. Epub 2014 May 5. PMID 24799476
- [Background] Kwon JH, Tanco K, Park JC, Wong A, Seo L, Liu D, Chisholm G, Williams J, Hui D, Bruera E. Frequency, Predictors, and Medical Record Documentation of Chemical Coping Among Advanced Cancer Patients. Oncologist. 2015 Jun;20(6):692-7. doi: 10.1634/theoncologist.2015-0012. Epub 2015 May 1. PMID 25933929
- [Background] Rudd RA, Seth P, David F, Scholl L. Increases in Drug and Opioid-Involved Overdose Deaths - United States, 2010-2015. MMWR Morb Mortal Wkly Rep. 2016 Dec 30;65(50-51):1445-1452. doi: 10.15585/mmwr.mm655051e1. PMID 28033313
- [Background] Le Merrer J, Becker JA, Befort K, Kieffer BL. Reward processing by the opioid system in the brain. Physiol Rev. 2009 Oct;89(4):1379-412. doi: 10.1152/physrev.00005.2009. PMID 19789384
- [Background] Kirsh KL, Jass C, Bennett DS, Hagen JE, Passik SD. Initial development of a survey tool to detect issues of chemical coping in chronic pain patients. Palliat Support Care. 2007 Sep;5(3):219-26. doi: 10.1017/s1478951507000387. PMID 17969825
- [Background] Vowles KE, McEntee ML, Julnes PS, Frohe T, Ney JP, van der Goes DN. Rates of opioid misuse, abuse, and addiction in chronic pain: a systematic review and data synthesis. Pain. 2015 Apr;156(4):569-576. doi: 10.1097/01.j.pain.0000460357.01998.f1. PMID 25785523
- [Background] Voon P, Karamouzian M, Kerr T. Chronic pain and opioid misuse: a review of reviews. Subst Abuse Treat Prev Policy. 2017 Aug 15;12(1):36. doi: 10.1186/s13011-017-0120-7. PMID 28810899
- [Background] Chou R, Turner JA, Devine EB, Hansen RN, Sullivan SD, Blazina I, Dana T, Bougatsos C, Deyo RA. The effectiveness and risks of long-term opioid therapy for chronic pain: a systematic review for a National Institutes of Health Pathways to Prevention Workshop. Ann Intern Med. 2015 Feb 17;162(4):276-86. doi: 10.7326/M14-2559. PMID 25581257
- [Background] Green CR, Anderson KO, Baker TA, Campbell LC, Decker S, Fillingim RB, Kalauokalani DA, Lasch KE, Myers C, Tait RC, Todd KH, Vallerand AH. The unequal burden of pain: confronting racial and ethnic disparities in pain. Pain Med. 2003 Sep;4(3):277-94. doi: 10.1046/j.1526-4637.2003.03034.x. PMID 12974827
- [Background] Bannan S, Danby A, Cowan D, Ashraf S, Martin PG. Low heparinization with heparin-bonded bypass circuits: is it a safe strategy? Ann Thorac Surg. 1997 Mar;63(3):663-8. doi: 10.1016/s0003-4975(96)01054-5. PMID 9066381
- [Background] Coleman JJ. The supply chain of medicinal controlled substances: addressing the Achilles heel of drug diversion. J Pain Palliat Care Pharmacother. 2012 Sep;26(3):233-50. doi: 10.3109/15360288.2012.703294. PMID 22973912